CLINICAL TRIAL: NCT05449041
Title: Validation of Bulbicam for Use on Patient Suffering From Glaucoma (GLA) and Cataract (CAT)
Brief Title: Bulbicam Validation on Glaucoma- and Cataract Patients
Status: Completed | Type: Observational
Sponsor: Meddoc (Other)
Responsible Party: Principal Investigator, Prof Stig Larsen, Research director, Meddoc
Other Study IDs: V2_OTH/GLA;CAT-I/2022
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma Eye; Cataract
Keywords: Bulbicam
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Glaucoma patients: Patients diagnosed with Glaucoma of both gender; passed the age of 18 years; without any other eye disease; suffering from other know serious disease but have a health situation in accordance with expectations related to the age.
  Interventions: Device: Bulbicam
- Glaucoma controlls: Gender- and age-matched controls to the Glaucoma patients, passed the age of 18 years without any eye diseases; not suffering from other know serious disease and have a health situation in accordance with expectations related to the age.
  Interventions: Device: Bulbicam
- Cateract patients: Patients diagnosed with Cataract of both gender; passed the age of 18 years; without any other eye disease; suffering from other know serious disease but have a health situation in accordance with expectations related to the age.
  Interventions: Device: Bulbicam
- Cataract controlls: Gender- and age-matched controls to the Cataract patients, passed the age of 18 years without any eye diseases; not suffering from other know serious disease and have a health situation in accordance with expectations related to the age.
  Interventions: Device: Bulbicam

INTERVENTIONS:
Device: Bulbicam — Measurement of eye pressure; Accuracy diagram; Contrast chart; Visual field, Pupil size
  Other Names: Standard eye examination devices

SUMMARY:
The aim is to investigate repeatability and stability of the six OTH-related Bulbicam tests in patients suffering from Glaucoma (GLA), b) Cataract (CAT) and matched healthy controls (HC).

The study population consists of the three subpopulations: 1) Patients suffering from GLA; 2) Patients suffering from CAT and 3) Gender- and age-matched HC without any eye diseases.

Bulbicam will be used in the study including six tests and the standard method will be used initially for measurements of "Visual Field" and "Pupil"

The study will be performed as a controlled, open, and non-randomized, stratified observational single center study. The stratification factors will be pathology and the degree of disease. Within each of the four strata, healthy matched controls related to gender and age (1:1) will be included.

The main variables will be the variables recorded at the six Bulbicam and the supporting variables will be recorded by the Standard (ST) investigation. The central variables related to Glaucoma will be the GAT and iCare pressure, "Seen /unseen "," Time until the given point is recorded as seen", "the light in decibel when the point is seen", X- and Y-coordinates and "Pupil diameter in mm".

The central variables related to cataract will be "Pupil diameter", "OCT RNFL ", "Seen /unseen "," Time until the given point is recorded as seen", "the light in decibel when the point is seen" and the X- and Y-coordinates.

Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. The Bulbicam examination will be performed twice a day with a rest period of one hour between each registration. This procedure will be repeated the following two days. All demographic data, social factors and history of disease will be recorded at screening.

Sixteen GLA-patients and 16 CAT-patients equally divided into two substrata will be recruited from the two participating hospitals. For each included patient, one gender- and age-matched HC will be recruited. In total 16 GLA-patients with 16 HC and 16 CAT-patients with 16 HC will be included in the study.

DETAILED DESCRIPTION:
Aim

* To investigate repeatability and stability of the six OTH-related Bulbicam tests in patients suffering from a) Glaucoma (GLA), b) Cataract (CAT) and matched healthy controls (HC).
* To compare Bulbicam and the standard method on measurements of Visual field and Pupil
* To contribute to establishment of normal range for GLA and CAT patients with different degrees in the disease development related to the Bulbicam tests.
* To contribute to establishment of normal range for a normal population without eye-disease related to the Bulbicam tests. Study population consists of the following three study populations: 1) Patients suffering from GLA of both genders above 18 years of age with different disease degree; 2) Patients suffering from CAT of both genders above 18 years of age with different disease degree; 3) Gender- and age-matched HC without any eye diseases.

Trial equipment: Bulbicam will be used in the study and the following six tests will be performed at each investigation: "Visual Field", "Ptosis", Dynamic Acuity", "Dynamic Contrast ", "Dark Adaption" and "Pupil". The standard method will be used initially for measurements of "Visual Field" and "Pupil"

Design:

The study will be performed as a controlled, open, and non-randomized, stratified observational single center study. The stratification factors will be pathology (GLA&CAT) and the degree of disease. Within each of the four strata, healthy matched controls related to gender and age (1:1) will be included. The degree of GLA is defined as follows:

1. Mild glaucoma
2. Moderate glaucoma
3. Severe glaucoma

The degree of CAT is defined as follows:

1. Cataract Nuclear Sclerosis - Grade 1
2. Cataract Nuclear Sclerosis - Grade 2

Higher grade cataracts are difficult to have occurred in Norway and thus excluded from this study.

For each included patient, a gender- and age-matched HV will be included. All included participants will perform Bulbicam eye-investigation twice at three flowing days with a rest period of at least one hour. Each investigation includes same six Bulbicam tests. The Standard method will only be performed once as the first investigation at day 1 for measurements of "Visual Field" and "Pupil".

Main variables will be the variables recorded at the six Bulbicam tests. Supporting Variables will be recorded by the Standard (ST) investigation for Glaucoma and Cataract.

The central variables related to Glaucoma will be the GAT and iCare pressure, "Seen /unseen "," Time until the given point is recorded as seen", "the light in decibel when the point is seen", X- and Y-coordinates and "Pupil diameter in mm". The central variables related to cataract will be "Pupil diameter", "OCT RNFL ", "Seen /unseen "," Time until the given point is recorded as seen", "the light in decibel when the point is seen" and the X- and Y-coordinates.

Study procedure:

Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. The Bulbicam examination will be performed twice a day with a rest period of one hour between each registration. This procedure will be repeated the following two days. All demographic data, social factors and history of disease will be recorded at screening. Additionally, the quality of life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be recorded initially as individual baseline values. The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for measuring and classifying the tolerability and toxicity at the end of each day of investigation.

Sample size:

Sixteen GLA-patients and 16 CAT-patients equally divided into two substrata will be recruited from the two participating hospitals. For each included patient, one gender- and age-matched HC will be recruited. In total 16 GLA-patients with 16 HC and 16 CAT-patients with 16 HC will be included in the study. All together the study will include 64 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with either Glaucoma or Cataract of both gender
* Passed the age of 18 years
* Without any other eye disease

Exclusion Criteria:

* Other visual disturbances and blindness
* Posterior Chamber Intraocular Lens (PCIOL)
* Physical or psychiatric disease, which may disturb the measuring procedure
* Patients who are not able to perform eye movements, so no full paresis of any ocular muscles
* Patients whose visual acuity is less than 0.1 in any eye, as these will not be able to focus on the test stimuli.
* Patients whose visible part of the eye is abnormal, such as subconjunctival hemorrhages or deformed pupils
* Patients whose pupils are not able to respond normally to dilation or contraction due to damaged nerves, mechanical damage of the pupil etc.
* With known alcoholic and drug dependency
* Not able to understand information.
* Not willing to give written consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study consists of the following three study populations: 1) Patients suffering from GLA of both genders above 18 years of age with different disease degree; 2) Patients suffering from CAT of both genders above 18 years of age with different disease degree; 3) Gender- and age-matched HC without any eye diseases.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
GAT | 0 hour
  Measurement of eye-pressure in mmHg
GAT | 1 hour
  Measurement of eye-pressure in mmHg
GAT | 24 hours
  Measurement of eye-pressure in mmHg
GAT | 25 hours
  Measurement of eye-pressure in mmHg
GAT | 36 hours
  Measurement of eye-pressure in mmHg
GAT | 37 hours
  Measurement of eye-pressure in mmHg
Visual Field | 0 hour
  Saccadic Reaction Time in ms
Visual Field | 1 hour
  Saccadic Reaction Time in ms
Visual Field | 24 hours
  Saccadic Reaction Time in ms
Visual Field | 25 hours
  Saccadic Reaction Time in ms
Visual Field | 36 hours
  Saccadic Reaction Time in ms
Visual Field | 37 hours
  Saccadic Reaction Time in ms
Ptosis | 0 hour
  MDR in mm
Ptosis | 1 hour
  MDR in mm
Ptosis | 24 hours
  MDR in mm
Ptosis | 25 hours
  MDR in mm
Ptosis | 36 hours
  MDR in mm
Ptosis | 37 hours
  MDR in mm
Dynamic Acuity | 0 hour
  Vision acuity in LogMar
Dynamic Acuity | 1 hour
  Vision acuity in LogMar
Dynamic Acuity | 24 hours
  Vision acuity in LogMar
Dynamic Acuity | 25 hours
  Vision acuity in LogMar
Dynamic Acuity | 36 hours
  Vision acuity in LogMar
Dynamic Acuity | 37 hours
  Vision acuity in LogMar
Dynamic Contrast | 0 hour
  Contrast sensitivity in LogCon
Dynamic Contrast | 1 hour
  Contrast sensitivity in LogCon
Dynamic Contrast | 24 hours
  Contrast sensitivity in LogCon
Dynamic Contrast | 25 hours
  Contrast sensitivity in LogCon
Dynamic Contrast | 36 hours
  Contrast sensitivity in LogCon
Dynamic Contrast | 37 hours
  Contrast sensitivity in LogCon
Dark Adaptation | 0 hour
  Fixed contrast; variable frequency in Hz
Dark Adaptation | 1 hour
  Fixed contrast; variable frequency in Hz
Dark Adaptation | 24 hours
  Fixed contrast; variable frequency in Hz
Dark Adaptation | 25 hours
  Fixed contrast; variable frequency in Hz
Dark Adaptation | 36 hours
  Fixed contrast; variable frequency in Hz
Dark Adaptation | 37 hours
  Fixed contrast; variable frequency in Hz
Pupil | 0 hour
  Diameter (mm)
Pupil | 1 hour
  Diameter (mm)
Pupil | 24 hours
  Diameter (mm)
Pupil | 25 hours
  Diameter (mm)
Pupil | 36 hours
  Diameter (mm)
Pupil | 37 hours
  Diameter (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Goran Petrovski, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Meddoc, Skjetten, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sverstad A, Helland-Hansen BA, Kristianslund O, Kolko M, Larsen SE, Petrovski G. Eye-tracking biomarkers for glaucoma based on saccadic reaction time: a controlled clinical study. Front Ophthalmol (Lausanne). 2025 Oct 16;5:1636911. doi: 10.3389/fopht.2025.1636911. eCollection 2025. PMID 41180014